CLINICAL TRIAL: NCT04101071
Title: Alternative Substrates in the Critically Ill Subject
Acronym: ASICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Bristol Royal Infirmary (Unknown); Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 266031
Record Dates: First submitted 2019-06-26; First posted 2019-09-24 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness
Keywords: Critical care; enteral feeding; nasogastric; ketogenic feed; feasibility
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: SIngle blinded, randomised, controlled feasibility study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modular ketogenic enteral feed (Experimental): Ketogenic enteral feed to be administered continuously for 10 days.
  Interventions: Other: Modular ketogenic feed
- Standard enteral feed (Active Comparator): Standard enteral feed to be administered continuously for 10 days.
  Interventions: Other: Standard feed

INTERVENTIONS:
Other: Modular ketogenic feed — Dietician prescribed, and consisting of Betaquik® (from Vitaflo, Nutritional company) to provide medium chain triglycerides), Renapro Shot® (protein), Maxijul® (carbohydrate) and multivitamins according to nutritional need (energy and protein requirements) based on clinical status of the participant. Ketogenic feed to be given continuously via nasogastric tube for 10 days
  Arms: Modular ketogenic enteral feed
Other: Standard feed — Standard Enteral feed. Dietician prescribed based on clinical status of the participant, as per individual Trust protocols. Standard feed to be given continuously via nasogastric tube for 10 days
  Arms: Standard enteral feed

SUMMARY:
The over-arching aim of this study is to investigate the feasibility of administrating alternative substrates to intensive care unit (ICU) patients. This includes reconstituting and administering a modular ketone-inducing (ketogenic) enteral feeding regimen to ICU patients; to show that this feed does increase blood ketones; and that it is feasible to collect the desired outcomes. This will allow us to determine in a subsequent randomised controlled trial whether this intervention improves ICU outcomes (including ICU-related muscle loss).

DETAILED DESCRIPTION:
Aggressive muscle wasting occurs early in critical illness, and is associated with a greater number of days on a ventilator, increased length of intensive care unit (ICU) and/or hospital stay, and subsequent functional impairment which may last years. Hospital care costs, and ongoing costs of community-based primary healthcare utilisation, are increased. No known interventions prevent this wasting.

Bioenergetic failure in critical illness and the potential for alternative substrate use:

Muscle protein synthesis is highly energy-dependent.The bioenergetic state of the critically-ill patient is compromised leading to decreased Adenosine Tri-Phosphate (ATP) synthesis. Alterations in mitochondrial function have been described repeatedly in the literature which, with other altered cellular processes, impair the utlilisation of metabolic substrates for ATP production.

Carbohydrate utilisation is impaired in critical illness, partly through impaired nuclear-to-membrane translocation of glucose transporter-4 and increased insulin resistance. Hypoxia signalling and inflammation block activity of pyruvate dehydrogenase by upregulation of pyruvate dehydrogenase kinase, increasing glucose availability thus driving pyruvate metabolism to lactate - the Pasteur effect.

The investigator's recently published data suggest that critical illness also impairs mitochondrial oxidation of fatty acids in skeletal muscle, and that the majority of lipids delivered in feed are not utilized for ATP production. This may be of clinical importance, given that lipids contribute 29-43% of the energy content of enteral, and 50% of parenteral, formulae. Lastly, oxidation of amino acids may produce ATP. However, this is not necessarily in the best interest of the patient: these amino acids are then no longer available for muscle protein synthesis. Further, most amino acid oxidation results in pyruvate production and therefore the same issues as those related to carbohydrate metabolism apply. Provision of a new metabolic substrate such as Ketone Bodies (KBs) may address these limitations.

Potential for Muscle Sparing Offered by Ketone Bodies:

During periods of starvation they may provide up to 50% of total body basal energy, enabling the high energy requirement of human brain to be met whilst sparing muscle. Additionally KBs may act as metabolic modulators, improving mitochondrial efficiency (also impaired by critical illness), and reducing reactive oxygen species and free radical formation. They also have anti-inflammatory effects (intramuscular inflammation is a driver of altered protein homeostasis, and anti-apoptotic activity. Together, these additional mechanistic effects may prove useful in ameliorating skeletal muscle wasting. Further, pilot data demonstrate a significant decrease in the plasma concentrations of beta-hydroxybutyrate and acetoacetate in early critical illness, consistent with increased KB uptake and utilisation early in critical illness.

Ketone bodies have diverse extra-mitochondrial metabolic effects. These include immune enhancement functions: specifically, to bacterial infection. Infection and inflammation are drivers of muscle wasting and amelioration of these may impact on this and other outcome measures. Thus, the critically ill patient may benefit from a ketogenic diet which have been used safely in other population groups, including healthy subjects the obese, and in patients with trauma, epilepsy, cardiovascular disease, Type-2 diabetes and Metabolic Diseases.

The objectives/aims are to:

1. Show that it is possible to recruit patients to receive a ketogenic feed
2. Show that it is possible for researchers to reconstitute the modular ketogenic feed on ICU.
3. Show that it is possible to administer ketogenic feed to ICU patients without ill effect.
4. Characterise the time-course of ketone generation (and related changes in related metabolic pathways) in response to the ketogenic feed.
5. Show that collection of outcome measures relevant for the subsequent substantive study will be feasible.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* due to receive enteral nutrition via nasogastric or nasojejunal tube as part of routine care
* mechanically ventilated and likely to remain so for >48 hours
* likely to remain on the ICU for >5 days
* likely to survive for at least 10 days and
* multi-organ failure (Sequential Organ Failure Assessment Score [SOFA] score >2 in 2 or more domains).

Exclusion Criteria:

* primary neuromyopathy or significant neurological impairment at the time of ICU admission that would preclude physical activity
* uni- or bilateral lower limb amputation
* requiring sole or supplemental parenteral nutrition
* need for specialist nutritional intervention
* patients with known inborn errors of metabolism
* participation in another clinical trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of patient recruitment; number eligible from screening | 15 months
  Number of patients screened
Feasibility of patient recruitment; percentage eligible from screening | 15 months
  Percentage of patients eligible for recruitment
Feasibility of patient recruitment; number from consent process | 15 months
  Number of eligible patients able to be consented to join the study
Feasibility of patient recruitment: percentage from consent process | 15 months
  Percentage of eligible patients able to be consented to join the study
Feasibility of patient retention during the 10 day study period: number of participants | 15 months
  Number of participants retained for the 10 day study; reasons for withdrawal analysed by descriptive statistics
Feasibility of patient retention during the 10 day study period; percentage of participants | 15 months
  Percentage of participants retained for the 10 day study; reasons for withdrawal analysed by descriptive statistics
Feasibility of provision of ketogenic feed: staff-completed questionnaire | 15 months
  Non-validated questionnaire to be completed by ICU bedside nurses and critical care research nurses within 2 weeks of recruitment completing. 12 questions will ask about ease of reconstituting and using the feed and any side effects encountered. Each question will be scored on a scale of 0-10 with 0 the worst/lowest score and 10 the best/highest score. The results for each question will be presented individually using descriptive statistics as mean +/- standard deviation, with a text description adding any comments received.
Incidence of Adverse Events/Serious Adverse Events, gastric intolerance, glucose variation | 15 months
  Percentage of days event occurred out of total possible days (mean +/- 95% confidence interval): pulmonary aspiration; vomiting, diarrhea (Bristol Stool Score T5-T7), prokinetics use, gastric residual volume >300mls; adverse blood glucose levels of >10.1mmol/l and <3.9mmol/l; Daily insulin use.
Coefficient of Glucose Variation (scored as mean/standard deviation) | 15 months
  Coefficient of Glucose Variation (scored as mean/standard deviation)
Timescale for the development and establishment of ketosis during 10 days of intervention or control feed; beta-hydroxybutyrate | 15 months
  Plasma levels of beta-hydroxybutyrate: mmol/l
Timescale for the development and establishment of ketosis during 10 days of intervention or control feed; acetoacetate | 15 months
  Plasma levels of acetoacetate mmol/l
Timescale for the development and establishment of ketosis during 10 days of intervention or control feed; pyruvate | 15 months
  Plasma levels of pyruvate mmol/l
Timescale for the development and establishment of ketosis during 10 days of intervention or control feed, fat | 15 months
  Plasma levels of fat (ratio of Medium Chain to Long Chain Triglyceride)
Timescale for the development and establishment of ketosis during 10 days of intervention or control feed, glucose | 15 months
  Plasma levels of glucose mmol/l
Timescale for the development and establishment of ketosis during 10 days of intervention or control feed, lactate | 15 months
  Plasma levels of lactate mmol/l

SECONDARY OUTCOMES:
Feasibility of data collection into electronic database from medical notes and nursing sheets as assessed by completion of >80% of available data: blood gases | 15 months
  Arterial Blood Gases, pH, PaO2 and PaCO2 in kPa
Feasibility of data collection into electronic database from medical notes and nursing sheets as assessed by completion of >80% of available data; biochemistry | 15 months
  Bicarbonate, Base Excess, Lactate, other biochemistry data in mmol/l
Feasibility of data collection into electronic database from medical notes and nursing sheets as assessed by completion of >80% of available data; haematology | 15 months
  Hematology data (Hb in g/l, White cell count and platelets in 10 to power of 9/l)
Feasibility of data collection into electronic database from medical notes and nursing sheets as assessed by completion of >80% of available data; bedside physiology | 15 months
  Bedside Physiology (BP, HR, SOFA score, Fluid Balance)
Feasibility of data collection into electronic database from medical notes and nursing sheets as assessed by completion of >80% of available data; nutritional data | 15 months
  Nutritional data (Protein g/kg/day and Energy kcal/kg/day
Feasibility of data collection into electronic database from medical notes and nursing sheets as assessed by completion of >80% of available data; Propofol | 15 months
  Propofol dose (mg/day)
Feasibility of performing quadriceps ultrasound scans: muscle mass | 15 months
  Ultrasound scans of rectus femoris part of quadriceps muscle as a measure of muscle mass
Feasibility of performing functional assessment at hospital discharge by Two- or Six-Minute Walk Test | 15 months
  Two minute or Six-Minute Walk Test (depending on patient capability) captures all the walking distance that a patient can demonstrate (in metres)
Feasibility of performing functional assessment at hospital discharge by Short Physical Performance Battery | 15 months
  Short Physical Performance Battery (scoring between 0-10; includes results of the gait speed, balance tests and chair stand)
Feasibility of performing functional assessment at hospital discharge by CPAx score | 15 months
  Chelsea Critical Care Physical Assessment Score (CPAx): scoring 0-5 in 10 domains
Feasibility of collecting metabolic data on ICU: indirect calorimetry | 15 months
  non-invasive metabolic data via indirect calorimetry on ICU
Feasibility of collecting follow-up data by telephone re quality of life: ED5Q survey | 18 months
  Use of ED5Q survey to determine health-related quality of life; scoring 1-5 in 5 domains, plus 1-100 in 1 domain
Feasibility of collecting follow-up data by telephone re job status: Questions on employment status | 18 months
  Questions on employment status (full-time: yes/no; part-time: yes/no)
Feasibility of collecting follow-up data from medical records: number of GP/nurse visits | 18 months
  Information on health care resource usage from number of GP/nurse visits during 12 months post-ICU and hospital discharge
Biochemical analysis of urine | 18 months
  To determine urinary concentrations of beta-hydroxybutyrate and total nitrogen (in mmol/l)
Biochemical analysis of plasma metabolites, beta-hydroxy butyrate, acetoacetate, leucine, and alanine (all measured in the same Arbitrary Units [AU]). | 18 months
  Investigation into beta-hydroxy butyrate, acetoacetate, leucine, and alanine (all measured in the same Arbitrary Units [AU]) by HPLC; NMR spectra will be phased, baseline corrected, zero filled and referenced prior to multivariate analysis. Multivariate techniques will include principal components analysis (PCA) and prediction and regression using partial least squared discriminant analysis (PLS-DA). Owing to the high variability expected in this data set, orthogonal projection to latent structures (OPLS) will be utilised to maximise the variation in the intervention under study. Given the high number of metabolites expected to be seen, statistical total correlation spectroscopy (STOCSY) will be utilised to detect endogenous responses.

CONTACTS AND LOCATIONS:
Overall Officials: Angela McNelly, PhD, Principal Investigator — Royal London Hospital
Locations (2):
- United Kingdom (2):
  - Bristol Royal Infirmary, Bristol
  - Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
(i) Where practicable, publicly funded research data should be made available for access, subject to such conditions as are necessary to ensure compliance with legal, data protection, ethical, confidentiality, intellectual property protection, and security/funder obligations.
  (ii) The rights of researchers to the exclusive use of research data that they generate as part of a well-defined research project will be protected up until the point of publication or public availability.
  (iii) Data arising from this research involving human subjects will be anonymised so that it will not be possible to identify any individuals. Where it appears inappropriate to make such data accessible, e.g. it might lead to identification of research subjects or because seeking consent would reduce the rate of participation in the research, the data will remain confidential.
  (iv) For research collaborations, any open access arrangements can only take place with the agreement of all research partners.
Supporting Information: Study Protocol
Time Frame: Data will be available once the primary publication is available. It will be available for a period of 10 years.
Access Criteria: Access is available for anyone who is able to provide a reasonable case for their access to the data.

REFERENCES:
- [Derived] McNelly A, Langan A, Bear DE, Page A, Martin T, Seidu F, Santos F, Rooney K, Liang K, Heales SJ, Baldwin T, Alldritt I, Crossland H, Atherton PJ, Wilkinson D, Montgomery H, Prowle J, Pearse R, Eaton S, Puthucheary ZA. A pilot study of alternative substrates in the critically Ill subject using a ketogenic feed. Nat Commun. 2023 Dec 15;14(1):8345. doi: 10.1038/s41467-023-42659-8. PMID 38102152